CLINICAL TRIAL: NCT04396106
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of AT-527 in Subjects With Moderate COVID-19
Brief Title: Safety and Efficacy of AT-527 in Subjects With Moderate Coronavirus Disease (COVID-19) in a Hospital Setting
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed out early due to evolving COVID-19 standard of care
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-03A-001
Record Dates: First submitted 2020-05-16; First posted 2020-05-20 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — AT-511

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AT-527 - 550 mg BID (Active Comparator): Part A
  Interventions: Drug: AT-527
- Placebo for 550 mg BID (Placebo Comparator): Part A
  Interventions: Other: Placebo
- AT-527 - 1100 mg BID (Active Comparator): Part B
  Interventions: Drug: AT-527
- Placebo for 1100 mg BID (Placebo Comparator): Part B
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AT-527 — One 550 mg tablet of AT-527 administered every ~12 hours (twice a day) for a total of 5 days
  Arms: AT-527 - 550 mg BID
Other: Placebo — One placebo tablet administered every ~12 hours (twice a day) for a total of 5 days
  Arms: Placebo for 550 mg BID
Drug: AT-527 — Two 550 mg tablets of AT-527 administered every ~12 hours (twice a day) for a total of 5 days
  Arms: AT-527 - 1100 mg BID
Other: Placebo — Two placebo tablets administered every ~12 hours (twice a day) for a total of 5 days
  Arms: Placebo for 1100 mg BID

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability, antiviral activity and efficacy of AT-527 in adult subjects ≥18 years of age with moderate COVID-19 and risk factors for poor outcomes (such as obesity (BMI>30), hypertension, diabetes or asthma). Eligible subjects will be randomized to blinded AT-527 (nucleotide analog) tablets or matching placebo tablets to be administered orally for 5 days. Part A will evaluate an AT-527 dose of 550 mg BID and Part B will evaluate a second dose of AT-527 (1100 mg BID). Local supportive standard of care (SOC) will be allowed for all subjects. Efficacy, antiviral activity and safety observations will be compared for treatment with active AT-527 tablets vs. placebo tablets.

ELIGIBILITY:
Key Inclusion Criteria:

* Hospitalized or in a hospital-affiliated confinement facility
* SARS-CoV-2 positive
* Initial COVID-19 symptom onset within 5 days prior to Screening
* SpO2 ≥ 93% on room air or requires ≤ 2L/min oxygen by nasal cannula or mask to maintain SpO2 ≥ 93%
* Must also have a history of at least one of the following known risk factors for poor outcomes: obesity (BMI>30), hypertension, diabetes or asthma.

Key Exclusion Criteria:

* Severe or critical COVID-19 illness: RR ≥30, HR ≥125, SpO2 <93% on room air or requires >2L/min oxygen by nasal cannula or mask to maintain SpO2 ≥93%, systolic blood pressure < 90 mm Hg, diastolic blood pressure < 60 mm Hg or PaO2/FiO2 <300
* Requires mechanical ventilation
* Lobar or segmental consolidation on chest imaging.
* Treatment with other drugs thought to possibly have activity against SARS-CoV-2
* ALT or AST > 5 x upper limit of normal (ULN)
* Female subject is pregnant or breastfeeding
* Has received or is expected to receive any dose of a SARS-CoV-2 vaccine before the Day 14 visit (Part B).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (14):
  - Atea Study Site, Scottsdale, Arizona
  - Atea Study Site, Davis, California
  - Atea Study Site, Los Angeles, California
  - Atea Study Site, Washington D.C., District of Columbia
  - Atea Study Site, Orlando, Florida
  - Atea Study Site, Atlanta, Georgia
  - Atea Study Site, Chicago, Illinois
  - Atea Study Site, Boston, Massachusetts
  - Atea Study Site, Butte, Montana
  - Atea Study Site, Charlotte, North Carolina
  - Atea Study Site, Cincinnati, Ohio
  - Atea Study Site, Columbus, Ohio
  - Atea Study Site, Charleston, South Carolina
  - Atea Study Site, Columbia, South Carolina
- Argentina (2):
  - Atea Study Site, Rosario
  - Atea Study Site, Vicente López
- Belgium (2):
  - Atea Study Site, Brussels
  - Atea Study Site, Mechelen
- Brazil (5):
  - Atea Study Site, Belo Horizonte
  - Atea Study Site, Brasília
  - Atea Study Site, Campo Largo
  - Atea Study Site, Porto Alegre
  - Atea Study Site, São Paulo
- Atea Study Site, Cairo, Egypt
- Atea Study Site, Chisinau, Moldova
- Atea Study Site, Bucharest, Romania
- South Africa (5):
  - Atea Study Site, Bloemfontein
  - Atea Study Site, Cape Town
  - Atea Study Site, Centurion
  - Atea Study Site, George
  - Atea Study Site, Worcester
- Spain (3):
  - Atea Study Site, Barcelona
  - Atea Study Site, Madrid
  - Atea Study Site, Pozuelo de Alarcón
- Ukraine (2):
  - Atea Study Site, Brovary
  - Atea Study Site, Kyiv

REFERENCES:
- [Derived] Horga A, Kuritzkes DR, Kowalczyk JJ, Pietropaolo K, Belanger B, Lin K, Perkins K, Hammond J. Phase II study of bemnifosbuvir in high-risk participants in a hospital setting with moderate COVID-19. Future Virol. 2023 Jun;18(8):489-500. doi: 10.2217/fvl-2023-0064. Epub 2023 Jun 23. PMID 38051993

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AT-527 - 550 mg BID | Placebo for 550 mg BID | AT-527 - 1100 mg BID | Placebo for 1100 mg BID
Started | 41 | 40 | 0 | 2
Completed | 37 | 37 | 0 | 1
Not Completed | 4 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | AT-527 - 550 mg BID | Placebo for 550 mg BID | AT-527 - 1100 mg BID | Placebo for 1100 mg BID | Total
Number analyzed (Participants) | 41 | 40 | 0 | 2 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.07) | 57.4 (8.33) |  | 33.5 (20.5) | 55.8 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 |  | 2 | 46
  Male | 22 | 15 |  | 0 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0
  Asian | 2 | 4 |  | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0
  Black or African American | 6 | 3 |  | 0 | 9
  White | 29 | 32 |  | 2 | 63
  More than one race | 2 | 1 |  | 0 | 3
  Unknown or Not Reported | 2 | 0 |  | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportions (Active vs. Placebo) of Subjects With Progressive Respiratory Insufficiency (PRI) on or Before Day 14.
Description: Progressive respiratory insufficiency defined as a ≥ 2-tier increase in respiratory support methods required to maintain satisfactory oxygenation (SpO2 ≥ 93%), using the 6-tier hierarchical scale of respiratory support methods, within the 14-day study period.
  Level 1:Normal oxygenation on room air (SpO2 ≥93), no need for supplemental O2 Level 2:Persistent hypoxemia on room air (SpO2 <93) with requirement for low-level supplemental O2 by nasal cannula/mask (up to 2L/min) to maintain SpO2 ≥93 Level 3:Requirement for higher levels of passive supplemental O2 by nasal cannula or mask (≥2 L/min) to maintain SpO2 ≥93 Level 4:Requirement for oxygenation by positive-pressure devices Level 5:Required invasive respiratory support (intubated mechanical ventilation or ECMO) Level 6:Death
Time Frame: Day 14
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | AT-527 - 550 mg BID | Placebo for 550 mg BID | AT-527 - 1100 mg BID | Placebo for 1100 mg BID
Number analyzed (Participants) | 41 | 40 | 0 | 2
Participants | 3 | 4 |  | 0
Statistical Analysis 1: Comparison: AT-527 - 550 mg BID vs Placebo for 550 mg BID; Test type: Other; p = 0.721, Cochran-Mantel-Haenszel

2. Secondary Outcome: Change From Baseline in Amount of SARS-CoV-2 Virus RNA by Nasopharyngeal Swab
Description: Change in the viral load as measured by swab of the upper part of the pharynx.
Time Frame: Through Day 14
Population: The modified intent-to-treat (mITT) analysis set included subjects who were randomized and treated and who had a positive SARS-CoV2 test result at baseline.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | AT-527 - 550 mg BID | Placebo for 550 mg BID | AT-527 - 1100 mg BID | Placebo for 1100 mg BID
Number analyzed (Participants) | 35 | 36 | 0 | 2
log10 copies/mL
  Change from baseline to Day 2: number analyzed (Participants) | 28 | 27 | 0 | 2
  Change from baseline to Day 2 | -0.55 (1.175) | -0.02 (1.838) |  | -1.37 (1.57)
  Change from baseline to Day 5: number analyzed (Participants) | 29 | 31 | 0 | 2
  Change from baseline to Day 5 | -1.00 (1.316) | -0.80 (1.853) |  | -2.51 (0.66)
  Change from baseline to Day 8: number analyzed (Participants) | 28 | 27 | 0 | 2
  Change from baseline to Day 8 | -1.64 (1.534) | -1.38 (1.281) |  | -3.78 (1.39)
  Change from baseline to Day 10: number analyzed (Participants) | 23 | 27 | 0 | 2
  Change from baseline to Day 10 | -1.72 (1.734) | -2.26 (1.452) |  | -4.78 (2.13)
  Change from baseline to Day 12: number analyzed (Participants) | 23 | 22 | 0 | 2
  Change from baseline to Day 12 | -2.13 (2.065) | -2.08 (1.584) |  | -4.78 (2.13)
  Change from baseline to Day 14: number analyzed (Participants) | 26 | 30 | 0 | 2
  Change from baseline to Day 14 | -2.61 (1.873) | -2.26 (1.747) |  | -4.13 (1.21)

ADVERSE EVENTS:
Time Frame: 28 days
Description: Treatment emergent adverse events (TEAEs) were defined as any adverse event that started or worsened in severity on or after the first dose of study drug.
Arm/Group | AT-527 - 550 mg BID | Placebo for 550 mg BID | AT-527 - 1100 mg BID | Placebo for 1100 mg BID
All-Cause Mortality (participants affected / at risk) | 0/40 | 2/40 | 0/0 | 1/2
Serious Adverse Events (participants affected / at risk) | 5/40 | 3/40 | 0/0 | 1/2
Other Adverse Events (participants affected / at risk) | 24/40 | 23/40 | 0/0 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AT-527 - 550 mg BID (N=40) | Placebo for 550 mg BID (N=40) | AT-527 - 1100 mg BID (N=0) | Placebo for 1100 mg BID (N=2)
Oxygen saturation decreased (Investigations) | 2 | 1 | NA | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | NA | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | NA | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | NA | 0
Haemodynamic instability (Vascular disorders) | 0 | 1 | NA | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | NA | 0
Pneumonia (Infections and infestations) | 0 | 1 | NA | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | NA | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AT-527 - 550 mg BID (N=40) | Placebo for 550 mg BID (N=40) | AT-527 - 1100 mg BID (N=0) | Placebo for 1100 mg BID (N=2)
Blood triglycerides increased (Investigations) | 6 | 6 | NA | 0
Alanine aminotransferase increased (Investigations) | 3 | 6 | NA | 0
Blood cholesterol increased (Investigations) | 5 | 2 | NA | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3 | NA | 0
Oxygen saturation decreased (Investigations) | 2 | 2 | NA | 0
Lipase increased (Investigations) | 1 | 2 | NA | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | NA | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 1 | NA | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | NA | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | NA | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | NA | 0
Injection site haemorrhage (General disorders) | 0 | 2 | NA | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | NA | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | NA | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | NA | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | NA | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 1
Pneumonia (Infections and infestations) | 0 | 2 | NA | 0

LIMITATIONS AND CAVEATS:
Study was prematurely discontinued. At the time of study discontinuation, only 2 subjects were enrolled in Part B and both received placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator may publish or present results pertaining to the PI's activities after the first publication of the multicentre clinical trial results, or 18 months after the clinical study database lock. Any such publications must be submitted for review by Sponsor before submission. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT04396106/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT04396106/SAP_001.pdf